CLINICAL TRIAL: NCT04904731
Title: Effects of Body Position on Diaphragmatic Activity in Patients Requiring Noninvasive Ventilation for Acute Respiratory Failure COVID-19 Related
Acronym: DiaCOVIDProne
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera di Perugia (Other)
Responsible Party: Principal Investigator, Prof Gianmaria Cammarota, Associate Clinical Professor, Azienda Ospedaliera di Perugia
Other Study IDs: 3658/20
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Noninvasive Ventlation; COVID-19 Respiratory Infection; Diaphragm Injury
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prone position — Patients were assisted in NIV in supine position that was switched in prone position for clinical purpouse

SUMMARY:
The present investigation aims to assess the diaphragmatic thickening fraction, reflecting the diaphragmatic activity, during supine (baseline) and at 1 hour following prone position in patients assisted through non invasive ventilation due to hypoxemic acute respiratory failure related to COVID-19. Also, the impact of lung aeration and comfort were ascertained in the same setting

DETAILED DESCRIPTION:
Primary aim is to asses the effects of body position on diaphragmatic thickening fraction (primary aim) and lung aeration and vital sign (secondary aims) in patents assisted via noninvasive ventilation (NIV) for hypoxemic acute respiratory failure (hARF) associated to COVID-19. All adult patients, admitted for hARF due to COVID-19 and requiring NIV were enrolled.

Diaphragmatic thickening fraction, lung aeration assessed through ultrasound, comfort, and grade of sedation-agitation as well as vital signs, i.e., peripheral oxygen saturation, blood pressure, and breathing pattern were monitored during noninvasive ventilation in supine and after 1 hour following the switch to prone position.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection,
* Age > 18 years,
* NIV application,
* ICU admission

Exclusion Criteria:

* Pregnancy,
* All the conditions contraindicating prone position and NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient, admitted to intensive care unit for hypoxemic acute respiratory failure associated to COVID-19 requiring NIV, who were subjected to prone position for clinical purpouse.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickening fraction | At baseline, in supine position
  The fraction of diaphragmatic thickness variations during respiratory cycle
Diaphragmatic thickening fraction | After 1 hour following prone position application
  The fraction of diaphragmatic thickness variations during respiratory cycle

SECONDARY OUTCOMES:
Lung aeration | At baseline, in supine position
  Lung aeration assessed through sonography
Peripheral oxygen saturation | At baseline, in supine position
  Reflects the grade of peripheral oxygenation
Lung aeration | after 1 hour following prone position application
  Lung aeration assessed through sonography
Peripheral oxygen saturation | after 1 hour following prone position application
  Reflects the grade of peripheral oxygenation

CONTACTS AND LOCATIONS:
Locations (1):
- Gianmaria Cammarota, Perugia, Umbria, Italy

IPD SHARING:
Plan to Share IPD: Undecided
single patients data on motivated request to principal investigator

REFERENCES:
- [Derived] Cammarota G, Rossi E, Vitali L, Simonte R, Sannipoli T, Anniciello F, Vetrugno L, Bignami E, Becattini C, Tesoro S, Azzolina D, Giacomucci A, Navalesi P, De Robertis E. Effect of awake prone position on diaphragmatic thickening fraction in patients assisted by noninvasive ventilation for hypoxemic acute respiratory failure related to novel coronavirus disease. Crit Care. 2021 Aug 24;25(1):305. doi: 10.1186/s13054-021-03735-x. PMID 34429131